CLINICAL TRIAL: NCT00863876
Title: Comparison of WaveLight Analyzer and Alcon LadarWave
Status: Completed | Type: Observational
Sponsor: WaveLight AG (Industry)
Responsible Party: Mr. Peter Riedel, WaveLight AG
Other Study IDs: S-388/2008
Record Dates: First submitted 2009-03-17; First posted 2009-03-18 (Estimated); Last update posted 2010-06-29 (Estimated); Status verified 2010-06

CONDITIONS: Healthy; Keratoconus
Keywords: wavefront measurements of the entire eye
MeSH Terms: conditions — Keratoconus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (9):
- 1: non-operated healthy eyes
- 2: eyes 1 months following LASIK
- 3: eyes 3-6 months following LASIK
- 4: eyes with spherical monofocal IOLs more than 3 months postop
- 5: eyes with aspherical monofocal IOLs more than 3 months postop
- 6: eyes with toric monofocal IOLs more than 3 months postop
- 7: eyes with diffractive multifocal IOLs more than 3 months postop
- 8: eyes with phakic IOLs more than 3 months postop
- 9: eyes with keratoconus

SUMMARY:
Comparison of repeated WaveLight Analyzer and Alcon LadarWave measurements in phakic and pseudophakic eyes.

ELIGIBILITY:
Inclusion Criteria:

* healthy eyes or eyes with the study conditions

Exclusion Criteria:

* age < 18, eye disorders other than mentioned above, participation in any other study,

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: healthy patients and patients following surgery, patients with keratoconus presenting for examination at the clinic
Sampling Method: Non-Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2009-03

CONTACTS AND LOCATIONS:
Locations (1):
- University of Heidelberg, Dept. of Ophthalmology, Heidelberg, Germany